CLINICAL TRIAL: NCT07358845
Title: Hematological Profiles of Preterm Infants: Can it be Effected by Antenatal Steroids?
Brief Title: Hematological Profiles of Preterm Infants and the Impact of Antenatal Steroids
Status: Completed | Type: Observational
Sponsor: Princess Anna Mazowiecka Hospital, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: ANS-HemProfiles
Record Dates: First submitted 2025-11-27; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Haematology
Keywords: haematological values; antenatal steroids; pregnancy; preterm infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 1.Optimal window (24hours-7days) group: Pregnant women who delivered 24 hours to 7 days after the last dose of antenatal steroids.
  Interventions: Drug: Antenatal Corticosteroid Exposure; Drug: Antenatal corticosteroids
- 2.Out-of-window (>7days) group: Pregnant women who delivered more than 7 days after antenatal steroid administration.
  Interventions: Drug: Antenatal Corticosteroid Exposure; Drug: Antenatal corticosteroids
- 3.Suboptimal (<24 hours) group: Pregnant women who delivered less than 24 hours after antenatal steroid administration.
  Interventions: Drug: Antenatal Corticosteroid Exposure; Drug: Antenatal corticosteroids
- 4.One-dose group: Pregnant women who received only the first dose of antenatal steroids before delivery.
  Interventions: Drug: Antenatal Corticosteroid Exposure; Drug: Antenatal corticosteroids
- 5.No steroids - lack of time: Pregnant women who did not receive antenatal steroids due to insufficient time before delivery.
- 6.No steroids - no recommendation: Pregnant women who did not receive antenatal steroids because therapy was not recommended.

INTERVENTIONS:
Drug: Antenatal Corticosteroid Exposure — Administration of ANS to pregnant women at risk of preterm delivery, according to standard clinical practice and existing obstetric guidelines. Corticosteroids were administered for fetal lung maturation. Exposure was categorized based on the interval between corticosteroid administration and delivery (24 hours to 7 days, less than 24 hours, more than 7 days), completeness of dosing (one dose only), or absence of exposure due to insufficient time before delivery or lack of clinical indication. This was an observational, exposure-based intervention.
  Groups: 1.Optimal window (24hours-7days) group; 2.Out-of-window (>7days) group; 3.Suboptimal (<24 hours) group; 4.One-dose group
Drug: Antenatal corticosteroids
  Groups: 1.Optimal window (24hours-7days) group; 2.Out-of-window (>7days) group; 3.Suboptimal (<24 hours) group; 4.One-dose group

SUMMARY:
The goal of this observational study is to investigate the impact of antenatal corticosteroids (ANS) administration on haematological parameters in premature infants born to women exposed to ANS.

The primary objective is to assess whether ANS administration in pregnant women during pregnancy alters haematological parameters in preterm neonates; The secondary objectives are: (1) to evaluate changes in haematological parameters in preterm infants in relation to the time interval between ANS administration and delivery, and (2) to assess alterations in haematological parameters according to different maternal ANS dosage regimens.

A total of 524 mother-infant pairs were included in the study. Participants were allocated into six groups based on the time interval between antenatal corticosteroid administration and delivery.

DETAILED DESCRIPTION:
Antenatal corticosteroids (ANS) have been widely used since 1972, when Liggins and Howie first demonstrated their beneficial effects on neonatal outcomes. Over time, the recognized benefits of ANS have extended beyond neonatal respiratory support in preterm infants. Current international guidelines recommend administering ANS to pregnant women at risk of imminent preterm delivery before 34 weeks of gestation. ANS therapy has been shown to reduce both morbidity and mortality among preterm neonates.

Glucocorticoid exposure promotes the maturation of multiple fetal organ systems, with a primary emphasis on accelerating lung development and reducing the risk of respiratory distress syndrome (RDS). The optimal therapeutic effect of ANS is observed within a window of 24 hours to 7 days following administration.

However, the potential adverse effects of corticosteroid therapy should not be overlooked and warrant careful consideration. First, corticosteroids may have negative effects on the developing brain, potentially leading to psychosomatic and neurodevelopmental disturbances, owing to the high density of glucocorticoid receptors in brain regions involved in behavioral regulation and endocrine control. Second, several studies have suggested that ANS may increase the risk of neonatal hypoglycemia and disrupt thyroid hormone homeostasis.

In addition, a study conducted by Romejko et al. demonstrated that ANS administration is associated with alterations in hematological parameters among women exposed to prenatal steroids.

Considering that anemia is a common condition among preterm infants, it is crucial to analyze additional factors that may influence hematological test results and complicate diagnostic evaluation. Therefore, reliable assessment of hematological parameters at birth is particularly important in this population.

The primary objective is to assess whether ANS administration in pregnant women during pregnancy alters haematological parameters in preterm neonates.

The secondary objectives are: (1) to evaluate changes in haematological parameters in preterm infants in relation to the time interval between ANS administration and delivery, and (2) to assess alterations in haematological parameters according to different maternal ANS dosage regimens.

ELIGIBILITY:
Inclusion Criteria:

* gestational age 24 weeks - <36 weeks

Exclusion Criteria:

* gestational age <24 and⩾36
* major congenital or chromosomal abnormalities
* intrauterine foetal demise
* women with active or suspected cancer
* women underwent surgery or chemotherapy during pregnancy
* women whose pregnancy was prematurely terminated due to maternal indications
* women who received ANS outside of our hospital
* lack of parental consent.

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We planned to recruit all consecutive pairs: pregnant women and their preterm infants admitted >24 and ≤ 36 weeks of gestation.
Sampling Method: Probability Sample
Enrollment: 1048 (Actual)
Dates: Start 2011-01-02 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2013-12-30 (Actual)

PRIMARY OUTCOMES:
Hemoglobin concentration [g/dl] in preterm infants <36 weeks of gestational age, measured in the first 24 hours of life | the first 24 hours of life
  Blood samples obtained within the first 24 hours of life; measured parameters will be compared between groups stratified by maternal ANS dosing regimen and interval between corticosteroid administration and delivery.
Hematocrit level [%] in preterm infants <36 weeks of gestational age, measured within the first 24 hours of life. | the first 24 hours of life
  Blood samples obtained within the first 24 hours of life; measured parameters will be compared between groups stratified by maternal ANS dosing regimen and interval between corticosteroid administration and delivery.
Red blood cell count (×10⁶/µL) in preterm infants <36 weeks of gestational age, measured within the first 24 hours of life. | the first 24 hours of life
  Blood samples obtained within the first 24 hours of life; measured parameters will be compared between groups stratified by maternal ANS dosing regimen and interval between corticosteroid administration and delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Romejko-Wolniewicz, Prof., M.D., Study Chair — Department of Obstetrics and Gynecology, Medical University of Warsaw, Poland
Locations (2):
- Poland (2):
  - Department of Obstetrics and Gynecology, Department of Neonatology and Neonatal Intensive Care, Warsaw, Medical University of Warsaw, Poland, Warsaw, Warsaw
  - Department of Obstetrics and Gynecology, Warsaw, Medical University of Warsaw, Poland, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be available. The study protocol will also be available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: november 2025-April 2026
Access Criteria: documents will be accessible to anyone who provides proposal following publication.

REFERENCES:
- [Background] Hasanbegovic E, Cengic N, Hasanbegovic S, Heljic J, Lutolli I, Begic E. Evaluation and Treatment of Anemia in Premature Infants. Med Arch. 2016 Dec;70(6):408-412. doi: 10.5455/medarh.2016.70.408-412. PMID 28210010
- [Background] Romejko-Wolniewicz E, Oleszczuk L, Zareba-Szczudlik J, Czajkowski K. Dosage regimen of antenatal steroids prior to preterm delivery and effects on maternal and neonatal outcomes. J Matern Fetal Neonatal Med. 2013 Feb;26(3):237-41. doi: 10.3109/14767058.2012.733758. Epub 2012 Oct 18. PMID 23035749
- [Background] Daskalakis G, Pergialiotis V, Domellof M, Ehrhardt H, Di Renzo GC, Koc E, Malamitsi-Puchner A, Kacerovsky M, Modi N, Shennan A, Ayres-de-Campos D, Gliozheni E, Rull K, Braun T, Beke A, Kosinska-Kaczynska K, Areia AL, Vladareanu S, Srsen TP, Schmitz T, Jacobsson B. European guidelines on perinatal care: corticosteroids for women at risk of preterm birth. J Matern Fetal Neonatal Med. 2023 Dec;36(1):2160628. doi: 10.1080/14767058.2022.2160628. PMID 36689999
- [Background] Battarbee AN, Ros ST, Esplin MS, Biggio J, Bukowski R, Parry S, Zhang H, Huang H, Andrews W, Saade G, Sadovsky Y, Reddy UM, Varner MW, Manuck TA; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Genomics and Proteomics Network for Preterm Birth Research (GPN-PBR). Optimal timing of antenatal corticosteroid administration and preterm neonatal and early childhood outcomes. Am J Obstet Gynecol MFM. 2020 Feb;2(1):100077. doi: 10.1016/j.ajogmf.2019.100077. Epub 2019 Dec 17. PMID 32905377